CLINICAL TRIAL: NCT01698827
Title: Replacement Gastrostomy Tubes: Technical and Clinical Comparison of Five Commercial Models
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Joel Faintuch, Associate Professor, Department of Gastroenterology, University of Sao Paulo
Other Study IDs: Gastrotubes5A
Record Dates: First submitted 2012-09-22; First posted 2012-10-03 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-09

CONDITIONS: Gastrostomy Tube Rupture; Gastrostomy Tube Durability; Gastrostomy Tube Convenience
Keywords: gastrostomy; tube; endoscopic; replacement; tube rupture; durability; tube loss; balloon rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Kangaroo: 20 patients managed by "Kangaroo" gastrostomy tubes. Patients will be submitted to initial screening and tube replacement, followed tube assessment visits every two months, till 6 months.
  Interventions: Other: Tube assessment visits
- Cook: 20 patients receiving "Wilson Cook" gastrostomy tubes.Patients will be submitted to initial screening and tube replacement, followed tube assessment visits every two months, till 6 months.
  Interventions: Other: Tube assessment visits
- Silmag: 20 patients managed by "Silmag" gastrostomy tubes.Patients will be submitted to initial screening and tube replacement, followed tube assessment visits every two months, till 6 months.
  Interventions: Other: Tube assessment visits
- Freka: 20 patients carrying "Freka" gastrostomy tubes.Patients will be submitted to initial screening and tube replacement, followed tube assessment visits every two months, till 6 months.
  Interventions: Other: Tube assessment visits
- Bard: 20 patients using the "Bard" gastrostomy tube. Patients will be submitted to initial screening and tube replacement, followed tube assessment visits every two months, till 6 months.
  Interventions: Other: Tube assessment visits

INTERVENTIONS:
Other: Tube assessment visits — Patients will return every 2 months for clinical questionnaire about leaks, obstructions or other dysfunctions of the tube. Objective tube examination for cracks, rupture, obstruction or dislodgement, along with replacement if necessary, will be carried out (total of 3 visits/6 months)

SUMMARY:
Multiple models of replacement tubes for percutaneous endoscopic gastrostomy are available in the market, however durability is variable. In a prospective randomized study, five commercial devices available in the market will be tested in 20 consecutive patients each. Tube performance will be observed during 6 months and durability will be assessed by Kaplan-Meier curves as well as Cox regression analysis.It is hypothesized that tube design and material will influence outcome.

DETAILED DESCRIPTION:
Multiple models of replacement tubes for percutaneous endoscopic gastrostomy are available in the market, however durability is variable. In a prospective randomized study, five commercial devices available in the market will be tested in 20 consecutive patients each,in patients submitted to long-term outpatient nutritional support. Tube performance will be observed during 6 months and durability will be assessed by Kaplan-Meier curves as well as Cox regression analysis.It is hypothesized that tube design and material will influence outcome.This study is important because tube dysfunction and unscheduled changes are expensive troubles that disrupt the nutritional protocol and are responsible for multiple inconveniences to the patient and the caretaker.

ELIGIBILITY:
Inclusion Criteria:

* Adults undergoing long-term home enteral nutrition via percutaneous endoscopic gastrostomy due to neurologic conditions or dysphagia.
* registered at the outpatient endoscopy service
* clinical stable and with the possibility of returning for scheduled visits
* expected duration of enteral feeding > 6 months

Exclusion Criteria:

* Sepsis,
* shock,
* coma,
* other types of digestive access (surgical gastrostomy, jejunostomy)
* terminal disease,
* lack of cooperation,
* refusal to participate in the protocol

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults on long-term nutritional care requiring prolonged gastrostomy feeding via percutaneous endoscopic gastrostomy
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Tube durability | 6 months
  Durability of the tube will be calculated as days in use till need for replacement, within the time frame of 6 months of observation. 180 days of continuous use will correspond to 100% durability, and 18 days of use as 10% durability.

SECONDARY OUTCOMES:
Tube rupture | 6 months
  Causes for replacement within the 6 months will be documented, with emphasis on tube or ballooon rupture

OTHER OUTCOMES:
Number of previous tube changes | 6 months
  Tube outcome will be analyzed in the light of number of previous tube changes in the patients (first tube/no previous change vs. patients on long-term treatment with multiple tube changes)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Faintuch, MD, PhD, Study Chair — Hospital das Clinicas, Sao Paulo, Brazil; Paulo Sakai, MD, PhD, Study Director — Hospital das Clinicas, Sao Paulo, Brazil; Emanuele L Villela, MD, Principal Investigator — Hospital das Clinicas, Sao Paulo, Brazil
Locations (2):
- Brazil (2):
  - Hospital das Clinicas- Central Institute ICHC- 9th Floor Rm 9077, São Paulo, São Paulo
  - Hospital das Clinicas, São Paulo, São Paulo

REFERENCES:
- [Background] Campoli P, Cardoso D, Turchi M, Mota O. Clinical trial: a randomized study comparing the durability of silicone and latex percutaneous endoscopic gastrostomy tubes. Dig Endosc. 2011 Apr;23(2):135-9. doi: 10.1111/j.1443-1661.2010.01051.x. Epub 2010 Dec 7. PMID 21429018
- [Derived] Villela EL, Sakai P, Almeida MR, Moura EG, Faintuch J. Endoscopic gastrostomy replacement tubes: long-term randomized trial with five silicone commercial models. Clin Nutr. 2014 Apr;33(2):221-5. doi: 10.1016/j.clnu.2013.04.015. Epub 2013 Apr 30. PMID 23672806